CLINICAL TRIAL: NCT00519649
Title: An Open, Phase IV, Single-group, Multicentre Study to Assess the Long-term Persistence of Antibodies Against Hepatitis B and the Immune Response to a Hepatitis B (HBV) Vaccine Challenge in Children Aged 7-8 Years of Age and Previously Vaccinated in Infancy With GSK Biologicals' HBV Vaccine (Engerix™-B).
Brief Title: Long-term Persistence of Immunity Against Hepatitis B in 7-8 Years Old Children After Hepatitis B Vaccination.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 110474
Record Dates: First submitted 2007-08-21; First posted 2007-08-22 (Estimated); Results first posted 2009-05-27 (Estimated); Last update posted 2018-08-17 (Actual); Status verified 2016-11

CONDITIONS: Hepatitis B Vaccine
Keywords: Hepatitis B vaccine; Challenge dose
MeSH Terms: conditions — Hepatitis B

ARMS (1):
- Group Engerix (Experimental): Subjects received a single challenge dose of Engerix™ (hepatitis-B [HBV] vaccine)
  Interventions: Biological: Engerix™-B Kinder

INTERVENTIONS:
Biological: Engerix™-B Kinder — Intramuscular injection, 1 dose

SUMMARY:
The purpose of this study is to assess the persistence of immunity to hepatitis B in children who received three consecutive doses of HBV vaccine (EngerixTM-B) in infancy. The Protocol Posting has been updated in order to comply with the FDA Amendment Act, Sep 2007.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who the investigator believes that their parents/guardians can and will comply with the requirements of the protocol.
* A male or female of 7 to 8 years of age (from and including the 7th birthday up to but excluding the 9th birthday) at the time of enrolment.
* With documented evidence of previous vaccination with three consecutive doses of Engerix™-B in Germany
* Written informed consent obtained from the parents or guardians of the subject at the time of enrolment.
* Healthy subjects as established by medical history and clinical examination before entering into the study.

Exclusion Criteria:

* Concurrently participating in another clinical study, at any time during the study period, in which the subject has been or will be exposed to an investigational or a non-investigational product
* Evidence of previous hepatitis B booster vaccination since administration of the third dose of Engerix™-B vaccine.
* History of or intercurrent hepatitis B disease.
* Hepatitis B vaccination at birth.
* Planned administration/administration of a vaccine not foreseen by the study protocol during the period starting from 30 days before HBV vaccine challenge and ending 30 days after.
* Administration of immunoglobulins and/or any blood products within the three months preceding HBV vaccine challenge or planned administration during the study period.
* Chronic administration (defined as more than 14 days) of immunosuppressants or other immune-modifying drugs within six months prior to the HBV vaccine challenge.
* Any confirmed or suspected immunosuppressive or immunodeficient condition, based on medical history and physical examination

Ages: 7 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 301 (Actual)
Dates: Start 2007-08-31; Primary Completion 2007-12-31 (Actual); Study Completion 2007-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (29):
- Germany (29):
  - GSK Investigational Site, Birkenfeld, Baden-Wurttemberg
  - GSK Investigational Site, Ettenheim, Baden-Wurttemberg
  - GSK Investigational Site, Heidelberg, Baden-Wurttemberg
  - GSK Investigational Site, Karlsruhe, Baden-Wurttemberg
  - GSK Investigational Site, Oberkirch, Baden-Wurttemberg
  - GSK Investigational Site, Oberstenfeld, Baden-Wurttemberg
  - GSK Investigational Site, Offenburg, Baden-Wurttemberg
  - GSK Investigational Site, Pforzheim, Baden-Wurttemberg
  - GSK Investigational Site, Stuttgart, Baden-Wurttemberg
  - GSK Investigational Site, Tuttlingen, Baden-Wurttemberg
  - GSK Investigational Site, Bindlach, Bavaria
  - GSK Investigational Site, Kaufering, Bavaria
  - GSK Investigational Site, Lohr, Bavaria
  - GSK Investigational Site, Munich, Bavaria
  - GSK Investigational Site, Tegernsee, Bavaria
  - GSK Investigational Site, Löhne, North Rhine-Westphalia
  - GSK Investigational Site, Minden, North Rhine-Westphalia
  - GSK Investigational Site, Münster, North Rhine-Westphalia
  - GSK Investigational Site, Porta Westfalica, North Rhine-Westphalia
  - GSK Investigational Site, Frankenthal, Rhineland-Palatinate
  - GSK Investigational Site, Mainz, Rhineland-Palatinate
  - GSK Investigational Site, Trier, Rhineland-Palatinate
  - GSK Investigational Site, Worms, Rhineland-Palatinate
  - GSK Investigational Site, Leipzig, Saxony
  - GSK Investigational Site, Bredstedt, Schleswig-Holstein
  - GSK Investigational Site, Flensburg, Schleswig-Holstein
  - GSK Investigational Site, Husum, Schleswig-Holstein
  - GSK Investigational Site, Kiel, Schleswig-Holstein
  - GSK Investigational Site, Berlin

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Derived] Behre U, Bleckmann G, Crasta PD, Leyssen M, Messier M, Jacquet JM, Hardt K. Long-term anti-HBs antibody persistence and immune memory in children and adolescents who received routine childhood hepatitis B vaccination. Hum Vaccin Immunother. 2012 Jun;8(6):813-8. doi: 10.4161/hv.19898. Epub 2012 Apr 17. PMID 22508412
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Study Protocol: 110474 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 110474 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 110474 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 110474 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 110474 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 110474 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 110474 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Recruitment Details: One additional subject, enrolled but not vaccinated, was not included in the number of subjects under "STARTED"
Period: Overall Study
Arm/Group | Group Engerix
Started | 300
Completed | 299
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Group Engerix
Number analyzed (Participants) | 300
Age, Continuous [Mean (Standard Deviation); unit: years] | 7.7 (0.46)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 136
  Male | 164

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Anti-hepatitis B Surface Antigen (HBs) Antibody Concentrations Above the Cut-off Value
Description: Anti-HBs antibody cut-off value assessed was 100 milli-international unit per milliliter (mIU/mL)
Time Frame: One month after the challenge dose of HBV vaccine
Population: Analysis was performed on the According-to-Protocol (ATP) cohort for analysis of immunogenicity
Measure: Count of Participants; unit: Participants
Arm/Group | Group Engerix
Number analyzed (Participants) | 280
Participants | 275

2. Secondary Outcome: Number of Participants With Anti-HBs Antibody Concentrations Above the Cut-off Value
Description: Anti-HBs antibody cut-off values assessed include 3.3, 10 and 100 mIU/mL
Time Frame: Before challenge dose of HBV vaccine
Population: Analysis was performed on subjects from the According-to-Protocol cohort for analysis of antibody persistence for whom serological results were available at pre-HBV vaccine challenge blood sampling time point
Measure: Count of Participants; unit: Participants
Arm/Group | Group Engerix
Number analyzed (Participants) | 282
Participants
  >= 3.3 mIU/mL | 261
  >= 10 mIU/mL | 235
  >= 100 mIU/mL | 104

3. Secondary Outcome: Number of Participants Reporting Solicited Local Symptoms
Description: Solicited local symptoms assessed include pain, redness and swelling
Time Frame: During the 4-day follow-up period after the challenge dose of HBV vaccine.
Measure: Count of Participants; unit: Participants
Arm/Group | Group Engerix
Number analyzed (Participants) | 299
Participants
  Pain | 89
  Redness | 81
  Swelling | 42

4. Secondary Outcome: Number of Participants Reporting Solicited General Symptoms
Description: Solicited general symptoms assessed include fatigue, fever, gastrointestinal symptoms, and headache
Time Frame: During the 4-day follow-up period after the challenge dose of HBV vaccine.
Measure: Count of Participants; unit: Participants
Arm/Group | Group Engerix
Number analyzed (Participants) | 299
Participants
  Fatigue | 44
  Fever (Axillary) | 9
  Gastrointestinal | 23
  Headache | 40

5. Secondary Outcome: Number of Participants Reporting Unsolicited Adverse Events
Description: An Adverse Event is any untoward medical occurrence in a clinical investigation subject, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product.
Time Frame: During the 31-day follow-up period after the challenge dose of HBV vaccine.
Measure: Count of Participants; unit: Participants
Arm/Group | Group Engerix
Number analyzed (Participants) | 300
Participants | 71

6. Secondary Outcome: Number of Participants Reporting Serious Adverse Events (SAE)
Description: An SAE is any untoward medical occurrence that:
  results in death, is life-threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, is a congenital anomaly/birth defect in the offspring of a study subject, or may evolve into one of the outcomes listed above.
Time Frame: After the challenge dose of HBV vaccine.
Measure: Count of Participants; unit: Participants
Arm/Group | Group Engerix
Number analyzed (Participants) | 300
Participants | 1

ADVERSE EVENTS:
Arm/Group | Group Engerix
All-Cause Mortality (participants affected / at risk) | 0/300
Serious Adverse Events (participants affected / at risk) | 1/300
Other Adverse Events (participants affected / at risk) | 159/300
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group Engerix (N=300)
Concussion (Injury, poisoning and procedural complications) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Group Engerix (N=300)
Pain (General disorders) | 89
Redness (General disorders) | 81
Swelling (General disorders) | 42
Fatigue (General disorders) | 44
Gastrointestinal (General disorders) | 23
Headache (General disorders) | 40

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.